CLINICAL TRIAL: NCT05670951
Title: A Multi-center, Double-Blind, Randomized, Two-Arm, Parallel-Group, Placebo Controlled Study to Assess the Efficacy and Safety of ELGN-2112 on Intestinal Malabsorption in Preterm Infants
Brief Title: Efficacy and Safety of ELGN-2112 on Intestinal Malabsorption in Preterm Infants
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Elgan Pharma Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FIT-PIV
Record Dates: First submitted 2023-01-02; First posted 2023-01-04 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Intestinal Malabsorption
MeSH Terms: conditions — Malabsorption Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ELGN-2112 (Active Comparator)
  Interventions: Drug: ELGN-2112
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ELGN-2112 — Human insulin [rDNA]
  Arms: ELGN-2112
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The study will evaluate the effect of ELGN-2112 on intestinal malabsorption in preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Male or female pre-term infant 26 and up to 32 weeks gestation. Gestational age matching (±2 weeks) between maternal dates and/or early antenatal ultrasound
* Birth weight ≥ 500g
* Singleton or twin birth

Exclusion Criteria:

-

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 360 (Estimated)
Dates: Start 2025-02-27 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
Numbers of days to achieve full enteral feeding | 28 days or discharge from hospital

CONTACTS AND LOCATIONS:
Locations (1):
- Laniado Hospital, Netanya, Israel